CLINICAL TRIAL: NCT00701896
Title: Smoking Cessation and the Natural History of HIV-Associated Emphysema
Brief Title: Smoking Cessation Using Motivational Therapy and Varenicline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Diaz (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Philip Diaz, Director, Pulmonary Rehabilitation Services; Medical Director, Respiratory Therapy; Associate Director, General Clinical Research Center, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007H0173; R01HL090313 (NIH)
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Smoking; HIV Infections
Keywords: HIV; Positive; Smokers; Varenicline
MeSH Terms: conditions — Smoking; HIV Infections | interventions — Varenicline; Nicotine Replacement Therapy; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Healthy Control - Non-smoking (Other): Healthy Control arm with 51 subjects who are HIV negative and do not smoke
  Interventions: Other: Biological Control
- Healthy Control - Smoker (Other): Healthy Control arm, includes 50 subjects who are HIV negative and are smokers.
  Interventions: Other: Biological Control
- HIV Smoking Cessation Arm (Active Comparator): Includes up to 365 subjects who are HIV positive and initiate smoking cessation
  Interventions: Drug: Varenicline tartrate; Drug: Nicotine Replacement Therapy
- Motivational Intervention (Experimental): Includes up to 100 subjects who are HIV positive, do not wish to quit smoking but are willing to undergo one-on-one Motivational Intervention
  Interventions: Behavioral: Motivational Interview

INTERVENTIONS:
Drug: Varenicline tartrate — 1 mMg tablet form; daily during week 1 (pre-quit week) followed by 1 mg twice daily for weeks 2-12.
  Other Names: Chantix
  Arms: HIV Smoking Cessation Arm
Drug: Nicotine Replacement Therapy — Nicotine gum and nicotine patch
  Arms: HIV Smoking Cessation Arm
Other: Biological Control — No treatment intervention only information and procedures.
  Arms: Healthy Control - Non-smoking; Healthy Control - Smoker
Behavioral: Motivational Interview — 60 minute one-on-one Interview
  Arms: Motivational Intervention

SUMMARY:
People that are infected with HIV appear to be especially susceptible to the adverse effects of cigarette smoking. The purpose of this study is to determine if quitting smoking by using a specialized smoking cessation treatment can prevent one from developing accelerated lung damage, particularly emphysema.

DETAILED DESCRIPTION:
HIV-infected smokers are at increased risk for life-threatening diseases, such as pneumonia. To date, very little is known about the tobacco consumption characteristics of this at-risk population of smokers, but it has been well documented that they are at high risk for smoking-related co-morbidities. In addition, few effective cessation strategies have been described in HIV-infected populations. A specialized smoking cessation that combines recommendations from an existing scientifically-valid clinical guideline with Motivational Interviewing a new pharmacotherapeutic agent, may be an effective mechanism to apply to this vulnerable population of smokers. This initial, efficacy investigation has the potential to guide future treatment and research pertaining to tobacco cessation, respiratory illness and HIV.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older;
2. diagnosis of HIV;
3. self-reported smoking on a daily basis;
4. provide informed written consent

Exclusion Criteria:

1. persons with active psychosis or impaired mental status as judged by the clinic staff and confirmed with a Mini-Mental Status Exam)
2. unable to understand spoken English
3. age less than 18 years.
4. pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2008-10-03 (Actual); Primary Completion 2013-04-20 (Actual); Study Completion 2013-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip T. Diaz, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Replacement Plus Motivational Interviewing: PLWH who smoke
  12 week intervention with telephone counseling plus:
  Nicotine Replacement Therapy: Nicotine gum (4 mg ad lib) and nicotine patch (21 mg)
- Varenicline Plus Motivational Interviewing: PLWH who smoke
  12 week intervention with telephone counseling plus:
  Varenicline tartrate: 0.5 mg daily days 1-3; 0.5 mg twice daily days 4-7; then 1.0 mg twice daily
Period: Overall Study
Arm/Group | Nicotine Replacement Plus Motivational Interviewing | Varenicline Plus Motivational Interviewing
Started | 143 (Includes those eligible but declined to participate) | 151 (Includes those eligible but declined to participate)
Completed | 110 | 118
Not Completed | 33 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Replacement Plus Motivational Interviewing | Varenicline Plus Motivational Interviewing | Total
Number analyzed (Participants) | 110 | 118 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 110 | 118 | 228
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 42.7 [20 to 63] | 42.8 [25 to 59] | 42.8 [20 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 93 | 101 | 194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 110 | 117 | 227
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 52 | 40 | 92
  White | 55 | 72 | 127
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 110 | 118 | 228

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Safety of Varenicline in PLWH Who Smoke
Description: To determine the safety and tolerability of varenicline compared to nicotine replacement
Time Frame: 3 months
Population: Three-month abstinence rates among participants who received NRT were compared with those who received varenicline. Although some participants stopped taking the pharmacotherapy, or switched from varenicline to NRT, for the analysis , they were kept in their initial group. Because treatment assignment was not random, inverse probability of treatment weighting (IPTW) adjustment was performed. A propensity score was estimated as the probability of receiving varenicline, given measured covariates
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Plus Motivational Interviewing | Varenicline Plus Motivational Interviewing
Number analyzed (Participants) | 110 | 118
Participants
  Nausea | 13 | 38
  Vomiting | 3 | 4
  Insomnia | 11 | 8
  Vivid dreams | 11 | 27
  Suicidal ideation | 0 | 1
  Depressed mood | 0 | 8
  Skin rash | 17 | 0

2. Secondary Outcome: To Determine the Efficacy of Varenicline for Smoking Cessation Among PLWH Who Smoke
Description: To compare biochemically confirmed tobacco abstinence rates among smokers living with HIV treated with nicotine replacement vs varenicline
Time Frame: 12 months
Population: Abstinence rates among participants who received NRT were compared with those who received varenicline. Although some participants stopped taking the pharmacotherapy, or switched from varenicline to NRT, for the analysis , they were kept in their initial group. Because treatment assignment was not random, inverse probability of treatment weighting (IPTW) adjustment was performed. A propensity score was estimated as the probability of receiving varenicline, given measured covariates
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Replacement Plus Motivational Interviewing | Varenicline Plus Motivational Interviewing
Number analyzed (Participants) | 110 | 118
Participants
  3 month biochemically confirmed abstinence rate | 13 | 30
  6 month biochemically confirmed abstinence rate | 5 | 19
  12 month biochemically confirmed abstinence rate | 4 | 18

ADVERSE EVENTS:
Arm/Group | Nicotine Replacement Plus Motivational Interviewing | Varenicline Plus Motivational Interviewing
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/110 | 1/118
Other Adverse Events (participants affected / at risk) | 56/110 | 94/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine Replacement Plus Motivational Interviewing (N=110) | Varenicline Plus Motivational Interviewing (N=118)
Suicidal Ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Replacement Plus Motivational Interviewing (N=110) | Varenicline Plus Motivational Interviewing (N=118)
Skin Rash (Skin and subcutaneous tissue disorders) | 17 (17) | 0 (0) — Skin rash
Skin redness (Skin and subcutaneous tissue disorders) | 6 | 0 (0)
Nausea (Gastrointestinal disorders) | 13 | 38
Insomnia (Psychiatric disorders) | 9 | 21
Vivid dreams (Psychiatric disorders) | 11 | 27
agitation (Psychiatric disorders) | 0 | 12
headache (Nervous system disorders) | 0 | 9
Constipation (Gastrointestinal disorders) | 0 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No